CLINICAL TRIAL: NCT03593434
Title: The Effect of Airway Clearance Therapy on Hyperpolarized 129Xenon MRI Compared With Lung Clearance Index and Spirometry in Cystic Fibrosis
Brief Title: Airway Clearance Therapy on Hyperpolarized 129Xenon and MRI
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason Woods, PhD, Director, Center for Pulmonary Medicine Imaging Research, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Other Study IDs: ACT and Xe MRI; 1R01HL131012-01A1 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-20 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hyperpolarized Xenon gas — This present study will utilize existing study visits for the NHLBI study, with patients opting-in to have all of the procedures performed twice, with an intervening ACT, during one their study visits.
  Other Names: 129Xenon

SUMMARY:
This is an observational cohort study building on an existing protocol at our institution recruiting CF patients who are 6-21 years old with one or two copies of the F508del CFTR mutation. That existing protocol seeks to enroll a total of 38 subjects; it includes three to four (three scheduled, with a fourth optional) study visits, with spirometry, LCI, UTE MRI, and 129Xe MRI being performed at each visit. This present study will utilize existing study visits for the NHLBI study, with a sub-set of 20 subjects opting-in to have all of the procedures performed twice, with an intervening ACT, during one of their study visits.

DETAILED DESCRIPTION:
This is an observational cohort study building on an existing protocol at our institution recruiting CF patients who are 6-21 years old with one or two copies of the F508del CFTR mutation. The existing protocol is funded by the NHLBI under R01-11863962 (PIs Woods, Clancy, and hereafter referred to as "the NHLBI study" for simplicity), and seeks to enroll a total of 38 subjects; it includes three to four (three scheduled, with a fourth optional) study visits, with spirometry, LCI, UTE MRI, and 129Xe MRI being performed at each visit. This present study will utilize existing study visits for the NHLBI study, with patients opting-in to have all of the procedures performed twice, with an intervening ACT, during one their study visits. The target enrollment is 20 subjects.

Airway clearance therapy (ACT) is used for treating cystic fibrosis (CF). It is known to impact measures of lung function, and while an increasing number of lung function measures are used in clinical trials, there has been no direct comparison of the effects of ACT across the different modalities. This study is actively investigating the relationship between different measures of lung function, comparing a spirometric measure (FEV1 percent-predicted) with measures of whole-lung ventilation (lung clearance index, or LCI) and regional assessments of both structure (with ultra-short echo time magnetic resonance imaging, or UTE MRI) and function (with hyperpolarized xenon, or 129Xe, MRI). Performing these assessments on CF patients will help to elucidate the relative sensitivity of each measure to intra-individual changes within the lung and will help guide the selection of lung function measures in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 through 21 years
* CFTR genotypes as specified in NHLBI study:

Two copies of the F508del CFTR mutation, OR Two non-functional CFTR mutations with one of them being F508del CFTR mutation

• Able to perform acceptable and repeatable spirometry

Exclusion Criteria:

* FEV1 percent predicted of <60%
* standard MRI exclusions (metal implants, claustrophobia)
* pregnancy

Ages: 6 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Male or female ages 6 through 21 with CF
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Effect of ACT on 129Xe MRI | one-day single study visit
  Quantify the effect of ACT on 129Xe MRI in ventilation defect percentage (%), in 20 children ages 6-21 years with CF

SECONDARY OUTCOMES:
Effect of ACT on spirometry | one-day single study visit
  Quantify the effect of ACT on spirometry in indexed values of FEV1, in percentage (%), in 20 children ages 6-21 years with CF
Effect of ACT on LCI | one-day single study visit
  Quantify the effect of ACT on lung clearance index (LCI) in LCI2.5 values, in 20 children ages 6-21 years with CF

OTHER OUTCOMES:
Structural changes on UTE MRI | one-day single study visit
  Describe the structural changes on UTE MRI that occur with airway clearance and correlate these with changes in spirometry and measures of ventilation heterogeneity

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided